CLINICAL TRIAL: NCT03171350
Title: A Prospective Multi-Centre Study of the Performance of the Ellume·Lab Group A Strep Test Versus Culture for the Rapid Detection of Group A Streptococcus in Participants With Acute Pharyngitis
Brief Title: Performance of Ellume·Lab Group A Strep Test Versus Culture for the Rapid Detection of Group A Streptococcus in Patients With Acute Pharyngitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-GAS-AUS-1701
Record Dates: First submitted 2017-05-28; First posted 2017-05-31 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Group A Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ellume.lab Group A Streptococcus Test (Experimental): ellume.lab Group A Streptococcus Test
  Interventions: Diagnostic Test: ellume.lab Group A Streptococcus Test

INTERVENTIONS:
Diagnostic Test: ellume.lab Group A Streptococcus Test — ellume.lab Group A Streptococcus Test is a rapid diagnostic test intended to be used as an aid in the diagnosis of Group A Streptococcus in symptomatic patients. The sample type used is a throat swab.

SUMMARY:
Participants who meet the eligibility criteria and who consent to participation or whose parents/legal guardian consent to their participation, will be enrolled in the study for a period of up to 14 days. Enrolment visit (Day 1) assessments for all participants will include the collection of throat swabs, testing by staff at the site using the ellume·lab Group A Strep Test and testing for Group A Streptococcus by a central laboratory using bacterial culture and polymerase chain reaction (PCR). All participants will be followed up with a phone assessment of adverse events between Days 2-14.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 3 years of age or older
* Must currently be presenting with symptoms characteristic of pharyngitis, possibly Group A Strep, including:

  * Acute onset of sore throat;
  * Fever ≥ 37.8° C (100° F) at presentation or history or parent/guardian-reported history of fever ≥ 37.8° C or feeling feverish within 24 hours of presentation and;
  * At least one of the following:

    * Red and swollen/inflamed tonsils;
    * Pharyngeal or tonsillar exudate; o Cervical lymphadenopathy
* ≤ 5 days from onset of signs and symptoms of pharyngitis
* Parent/legal guardian of Participants < 18 years of age capable and willing to give informed consent
* Participants ≥18 years of age capable and willing to give informed consent

Exclusion Criteria:

* Participants < 3 years of age
* Participants undergoing treatment with antibiotics, or those who have undergone treatment with antibiotics for current episode of pharyngitis
* Participants who have pharyngitis with clinical features that suggest a viral etiology such as, cough, runny nose, upper respiratory symptoms, and/or oral ulcers
* Currently enrolled in another clinical trial or used any investigational device within 30 days preceding informed consent
* Participants 18 years of age or older unable to understand English and consent to participation
* Parent/legal guardian of Participants < 18 years of age unable to understand English and consent to participation of child

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to bacterial culture | 1 week
The specificity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to bacterial culture | 1 week
The overall agreement between the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab and results from bacterial culture | 1 week

SECONDARY OUTCOMES:
The sensitivity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to PCR | 1 week
The specificity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using throat swab as compared to PCR | 1 week
The overall agreement between the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab and results from PCR | 1 week
Ease of use as assessed by operator questionnaire. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Glen Mulhall, Principal Investigator — University of the Sunshine Coast Clinical Trials Centre
Locations (8):
- Australia (8):
  - Ochre Health Medical Centre, Casey, Australian Capital Territory
  - Forbes Medical Centre, Forbes, New South Wales
  - Paratus Clinical Wyong Clinic, North Sydney, New South Wales
  - Mingara Medical, Tumbi Vmbi, New South Wales
  - Wamberal Surgery, Wamberal, New South Wales
  - Paratus Clinical Wyoming Clinic, Wyoming, New South Wales
  - USC Clinical Trials Centre, Maroochydore, Queensland
  - Griffith University Clinical Trial Unit, Southport, Queensland

IPD SHARING:
Plan to Share IPD: No